CLINICAL TRIAL: NCT03262454
Title: Sequential Hypofractionated Radiotherapy Followed by Anti-PD-L1 Atezolizumab for Recurrent or Refractory Small Cell Lung Cancer
Brief Title: Sequential Hypofractionated Radiotherapy Followed by Anti-PD-L1 Atezolizumab for SCLC
Acronym: Atezolizumab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Roche Korea co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Ji-youn Han, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2017-0229; ML39728 (Other Grant/Funding Number: Roche Korea Ltd)
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Small Cell Lung Cancer Recurrent
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventions (Experimental): Atezolizumab
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Patients undergo hypofractionated radiation therapy with 24 Gy over 4 fractions in days 1-4 of 1st cycle of atezolimumab and receive Atezolizumab 1200 mg fixed dose via intravenous on day 1 of each 3-week cycle until disease progression or unacceptable toxicity occurs.
  Other Names: Tecentriq

SUMMARY:
The investigators hypothesized that local radiation therapy can enhance the effect of anti-PD-L1 monoclonal antibody through priming T-cell effector function against cancer cells. Described as above, The investigators concluded that modest dose of radiation to local site prior to immunotherapy is the best to enhance T-cell-mediated immunity. Accordingly, The investigators will investigate the combining effect of hypofractionated-sublethal dose of radiation therapy followed by anti-PD-L1 monoclonal antibody, atezolizumab, for SCLC patients who are recurrent or refractory for initial platinum-based chemotherapy

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC), accounting for 10% of all lung cancers (Torre et al., 2015), shows poor outcomes with 7-10 months of median survival in advanced cases (Jett et al., 2013). Despite novel treatment strategies including targeted therapy and immunotherapy for non-small cell lung cancer (NSCLC) have been introduced, the treatment options for SCLC still remain limited. Many clinical trials, which tested the efficacy of molecular targeted agents for SCLC, failed to show clinical benefit compared with conventional platinum-based chemotherapy (Koinis et al., 2016). Nevertheless, recent studies demonstrated that immunotherapy using anti-CTLA-4 or anti-PD1 monoclonal antibody can be novel therapeutic strategies for SCLC (Ott et al., 2015; Reck et al., 2013; SJ et al., 2015).

In recent years, many studies have shown that radiation therapy can be a useful treatment as a combining treatment with immunotherapy. The abscopal effect refers to the ability of radiation delivered radiation delivered to a local site to treat the other diseases outside radiation field (Tang et al., 2014). A recent study described that abscopal effect was observed in a malignant melanoma patient treated with CTLA4 antagonist and radiotherapy (Postow et al., 2012). Moreover, an animal study presented that blockade of PD-L1 and ionizing radiation showed synergism (Deng et al., 2014). Based on these emerging evidences, the investigators hypothesized that local radiation therapy can enhance the effect of anti-PD-L1 monoclonal antibody through increasing T-cell effector function against tumors. Atezolizumab, which is a humanized anti-PD-L1 monoclonal antibody, act as an inhibitor the interaction between PD-L1 and PD-1, and eventually restore suppressed T-cell immunity leading elimination of cancer cells. In this study, the investigators will investigate the combining effect of hypofractionated-sublethal dose of radiation therapy followed by anti-PD-L1 monoclonal antibody, atezolizumab, for SCLC patients who are recurrent or refractory for initial platinum-based chemotherapy.

Based on these emerging evidences, the investigators hypothesized that local radiation therapy can enhance the effect of anti-PD-L1 monoclonal antibody through priming T-cell effector function against cancer cells. Described as above, the investigators concluded that modest dose of radiation to local site prior to immunotherapy is the best to enhance T-cell-mediated immunity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 18 years or older
2. Histologically confirmed SCLC and available tumor tissues for PD-L1 staining
3. Progression during or after platinum-based chemotherapy.
4. At least one target tumor lesion that has not been irradiated within the past three months and that can accurately be measured in at least one dimension with longest diameter
5. Life expectancy of at least three months
6. Performance status of 0, 1, 2 on the ECOG criteria
7. Adequate hematologic and end-organ function, Patients may be transfused or receive erythropoietic treatment to meet this criterion.
8. Patient has given written informed consent which must be consistent with the International Conference on Harmonization - Good Clinical Practice (ICH-GCP) and local legislation

Exclusion Criteria:

1. Previous therapy with anti-PD-1 or -PD-L1 inhibitors
2. Persistence of clinically relevant therapy related toxicities from previous chemotherapy and/or radiotherapy
3. Chemotherapy, treatment with tyrosine kinase inhibitors, or radiotherapy (except for brain and extremities) within the past 3 weeks prior to treatment with the trial drug i.e., the minimum time elapsed since the last anticancer therapy and the first radiotherapy must be 3 weeks
4. Treatment with other investigational drugs or treatment in another clinical trial within the past three weeks before start of therapy or concomitantly with this trial
5. Concomitant yellow fever vaccination
6. Active or untreated CNS metastases as determined by CT or MRI evaluation during screening and prior radiographic assessments
7. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for 2 weeks prior to randomization
8. Leptomeningeal disease
9. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
10. Uncontrolled tumor-related pain
11. Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
12. Significant cardiovascular diseases (i.e., hypertension not controlled by medical therapy, unstable angina, history of myocardial infarction within the past 12 months, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion)
13. Proteinuria CTCAE grade 2 or greater
14. Significant weight loss (> 10 %) within the past 6 weeks prior to treatment in the present trial
15. Current peripheral neuropathy ≥ CTCAE(version4.0) Grade 2 except due to trauma
16. Major injuries and/or surgery with incomplete wound healing within the past ten days prior to enrollment
17. Serious infections requiring systemic antibiotic (e.g. antiviral, antimicrobial, antifungal) therapy
18. Active hepatitis C and/or B infection
19. Known human immunodeficiency virus (HIV) seropositivity
20. Serious illness or concomitant non-oncological disease such as neurologic-,psychiatric-, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
21. Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least 5 months after end of active therapy
22. Pregnancy or breast feeding
23. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
24. Patients unable to comply with the protocol
25. Active alcohol or drug abuse
26. Other malignancy within the past three years other than basal cell skin cancer or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2023-02-23 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, and average of 1 years
  Objective Response rate using RECIST v1.1

SECONDARY OUTCOMES:
PFS | From date of enroll until the date of first documented progression or date of death from any cause, whichever came first, assessed up to at least 12 months
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea